CLINICAL TRIAL: NCT04605601
Title: The Effects of Virtual Reality on Upper Extremity in Patients With Obstetric Brachial Plexus Injury
Brief Title: The Effects of Virtual Reality Patients With Obstetric Brachial Plexus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Atıcı (Other)
Responsible Party: Sponsor-Investigator, Emine Atıcı, Physiotherapist, PhD, Okan University
Organization: Okan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-10-22; First posted 2020-10-28 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Obstetric Brachial Plexus Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental)
  Interventions: Other: Virtual reality treatment
- Control Group (Other)
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: Virtual reality treatment — Tennis, boxing, and baseball games of the Wii Sports package sre used for activating the upper extremity functions of the patients. In the tennis game, patients represent people holding rackets.
  Arms: Study Group
Other: conventional physiotherapy — As the conventional physiotherapy, neuromuscular electrical stimulation and strengthening exercises for the deltoid, infraspinatus, triceps, biceps, supinator, and wrist extensor muscles, and passive, active, active assistive joint Rage of Motion, and stretching exercises for the shoulder, elbow and wrist joints are applied to the patients in the standardized program for the upper extremity in 10 repetitions.
  Arms: Control Group

SUMMARY:
Obstetric brachial plexus injury is the flask paralysis of the arm, which emerges from a difficult birth. This results from the damage to the nerves from the C5 cervical root to T1. Following brachial plexus injury, movement impairment, a decrease in the joint range of motion, muscle contractures, motor disorders related to muscle weakness, and the loss of functional movements are commonly observed. Many rehabilitation programs for the upper extremity aim at developing functional improvement in addition to increasing the active range of motion of the related limb in children with Obstetric brachial plexus injury. Obstetric brachial plexus injury treatment includes both conservative and surgical interventions. The first intervention in all the Obstetric brachial plexus injury cases is conservative. In recent years, supporting the treatment with virtual reality exercises in addition to the conventional brachial plexus rehabilitation is a method being tested. The use of virtual reality treatment in physiotherapy and rehabilitation has substantially increased within the last 6-7 years. Virtual reality is a method that enables working with task-based techniques by creating stimulating and entertaining environments and especially using children's interest and motivation. Nintendo Wii, which is used in the virtual reality treatment, is a device that can be controlled wirelessly, consists of a system console, remote control for activity control, and a sensor perceiving the change in movements, and a display screen, and gives the opportunity to work with the person individually. The aim of this study is to investigate the effects of the conventional physiotherapy approach and virtual reality applications with Nintendo Wii, applied additionally in this study, on upper extremity functions in children with obstetric brachial plexus injury. They can directly be mentioned as the effects on muscle strength, normal joint range of motion, and functionality.

ELIGIBILITY:
Inclusion Criteria:

* undergone primary or -if available- secondary surgery at least 6 months before
* Being between the ages of 5-13
* be affected by the C5-C6 (upper truncus)

Exclusion Criteria:

* Patients with severe cognitive functional disorder
* Patients with cognitive functions inadequate for communication
* Patients with any neurological problems
* Patients who have a contracture preventing the upper extremity joints from performing activities

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Active Movement Scale | 4 weeks
  The Active Movement Scale, developed by Clarke and Curtis, was specifically developed for children with neonatal (between the ages of 0-1) obstetric brachial plexus palsy, and it was developed as a scoring system that consists of eight sequential steps and can numerically measure the upper extremity strength. It allows for scoring against gravity and in positions with the elimination of gravity in the score interval of "0-7" for 15 joint movements in the upper extremity. While scoring the joint movement in the position with the elimination of gravity in the score interval of "0-4", the same movement is repeated in children who can receive "4" against gravity, and the score interval of "5-7" is evaluated. The advantage of the Active Movement Scale is its frequent use in this field and its applicability until adolescence.
Mallet Scoring System | 4 weeks
  Another way of evaluating children with Obstetric Brachial Plexus Injury is the Mallet Scoring System. The Mallet Scoring System is often used for evaluating the shoulder function. Since the child needs to perform the desired movements actively, it is more appropriate to use this scale in children older than 3-4 years of age. The patient is expected to actively perform 5 different shoulder movements such as shoulder abduction, moving the hand towards the head, back, and mouth. Each movement is assessed between 1 and 5 (1st degree: Total paralysis, 5th degree: normal joint shoulder movement).
Normal Joint Range of Motion | 4 weeks
  In our study, the active and passive shoulder flexion, abduction and internal-external rotation, elbow flexion, forearm supination-pronation, and wrist flexion-extension of all the patients on the affected side are evaluated in the supine position before and after the treatment. The limited movements of the upper extremity were measured using a digital goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Emine Atıcı, Tuzla, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No